CLINICAL TRIAL: NCT04490174
Title: Serological Surveillance for COVID-19 in Central North Carolina
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200143; 20-E-0143
Record Dates: First submitted 2020-07-28; First posted 2020-07-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Natural History
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants: Healthy adults without a current active COVID-19 infection or current symptoms consistent with COVID-19 at the first clinic visit

SUMMARY:
Background:

The SARS-CoV-2 virus has caused a pandemic. Little is known about the virus, so data is needed to form an effective public health response. Researchers want to count how many people have been exposed to COVID-19, learn about symptoms, and find out how many antibodies to the SARS-CoV-2 virus a person may have in their blood over 1 year. This data could affect the response to current and future pandemics.

Objective:

To learn how many people from a sampling of adults in North Carolina develop antibodies to the SARS-CoV-2 virus over 1 year.

Eligibility:

Healthy people age 18 and older who do not currently have COVID-19

Design:

Participants will be screened with questions about their health.

Participants will have five 30-minute visits at the Clinical Research Unit. At each visit, they will have blood drawn to see if they have SARS-CoV-2 antibodies.

If the test result is positive for antibodies, the participant will be tested to see if they currently have COVID-19. For this, a nasal or throat swab will be done, or saliva will be collected. They may do this test at the same visit as the blood draw, or they may schedule an extra visit.

Around the time of their study visits, participants will take an online survey about themselves, their health, and COVID-19. It takes 10 minutes to complete. Every week for 52 weeks, they will also take a brief online survey about their symptoms. It takes 2 minutes to complete. They will be emailed a link to log in and fill out the surveys on a secure website.

Participation will last for 1 year.

DETAILED DESCRIPTION:
It has been demonstrated that respiratory virus outbreaks and pandemics, such as influenza, SARS, MERS, and now the newly emerged SARS-CoV-2 virus, have a major impact on morbidity and mortality worldwide, as well as having devastating global economic and societal impact. During these outbreaks it is critical to gain a rapid understanding of the exposures and immunity in the general population. Identifying exposures can be accomplished through analysis of serum during an outbreak to identify those with specific antibodies to the pathogen.The knowledge of the level of exposures could greatly impact the response to current and future pandemics.

This study is a prospective, longitudinal, observational, single-center, exploratory, natural history study to collect samples and data from individuals to identify the presence and rate of development of anti-SARS-CoV-2 antibodies in North Carolina.

Objectives: Primary Objective:

To characterize the proportion of people with detectable antibodies to SARS-CoV-2 from a sampling of adults in North Carolina.

Exploratory Objectives:

* To identify the incidence of newly detectable antibodies to SARS-CoV-2 in the recruited cohort of adults in North Carolina over 12 months after enrollment
* To identify the rate of asymptomatic carriers of SARS-CoV-2 (PCR positive) among participants with detectable antibodies to SARS-CoV-2
* To associate presence or absence of detectable antibodies to SARS-CoV-2 with respiratory symptoms and future diagnosis with COVID-19
* To determine the natural history of antibody titers among the participants who are found to have detectable antibodies
* To associate demographic and medical factors with incidence of newly detectable antibodies to SARS-CoV-2

Endpoints: Primary Endpoint:

- Detection of Anti-SARS-CoV-2 antibodies by ELISA Assay Algorithm

Exploratory Endpoints:

1. SARS-CoV-2 PCR of nasal swabs and correlation with serology
2. Clinical questionnaire data and correlation with serology and PCR

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male and females
2. greater than or equal to 18 years of age
3. Able to read and speak English
4. Ability to provide informed consent
5. Able to travel to study visits at the NIEHS CRU for required study visits
6. Stated willingness to comply with all study procedures and availability for the duration of the study

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Current symptoms consistent with COVID-19 infection at the point of Antibody Visit 1
2. Inability to provide a blood sample
3. Current pregnancy or lactation, by participant verbal confirmation.
4. Any condition that, in the investigator's opinion, places the participant at undue risk for complications associated with required study procedures.
5. Not willing to have blood samples stored for future research

Participants who have Limited English Proficiency will be excluded from the study because the informed consent form is only available in English. The study documents (Demographic and Health Assessment Questionnaire, and Weekly Symptom Questionnaire) and FDA Fact Sheets for Tests with Emergency Use Authorization are only available in English.

Decisionally impaired adults and prisoners will be excluded due to the inability to complete necessary study procedures. Adults who become prisoners or decisionally impaired while on study will be withdrawn.

Pregnant women are excluded due to the need to have participants venture out during the COVID-19 pandemic. Women who become pregnant during the study will be withdrawn.

Children will be excluded from enrolling in this study as immunity in children is different than

adults and we are focusing on adult immunity and in this trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults >18 years age without a current active COVID-19 infection or current symptoms consistent with COVID-19 within Central North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Anti-SARS-COV-2 antibodies | Day1, months 3, 6, 9, 12
  Proportion of people with detectable Anti-SARS-COV-2 antibodies

SECONDARY OUTCOMES:
Positive SARS-CoV-2 PCR | Day1, months 3, 6, 9, 12
  To identify the rate of asymptomatic carriers of SARS-CoV-2 (PCR positive) among participants with detectable antibodies to SARS-CoV-2
Detection of Anti-SARS-CoV-2 antibodies by ELISA Assay Algorithm | Day1, months 3, 6, 9, 12
  To identify the incidence of newly detectable antibodies to SARS-CoV-2 in the recruited cohort of adults in North Carolina over 12 months after enrollment
Detection of Anti-SARS-CoV-2 antibodies by ELISA Assay Algorithm | Day1, months 3, 6, 9, 12
  To determine the natural history of antibody titers among the participants who are found to have detectable antibodies
Clinical questionnaires and ELISA antibody testing results | Day1, months 3, 6, 9, 12
  To associate presence or absence of detectable antibodies to SARS-CoV-2 with respiratory symptoms and future diagnosis with COVID-19
Clinical questionnaires and ELISA antibody testing results | Day1, months 3, 6, 9, 12
  To associate demographic and medical factors with incidence of newly detectable antibodies to SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Garantziotis, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Background] Tandon PN. COVID-19: Impact on health of people & wealth of nations. Indian J Med Res. 2020 Feb & Mar;151(2 & 3):121-123. doi: 10.4103/ijmr.IJMR_664_20. No abstract available. PMID 32202260
- [Background] Dong L, Bouey J. Public Mental Health Crisis during COVID-19 Pandemic, China. Emerg Infect Dis. 2020 Jul;26(7):1616-1618. doi: 10.3201/eid2607.200407. Epub 2020 Jun 21. PMID 32202993
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-E-0143.html